CLINICAL TRIAL: NCT06926010
Title: Effect of a Predictive Hemodynamic Approach on the Stump Pressure During Carotid Endoartectomy: a Randomized Controlled Trial
Brief Title: Hemodynamic Monitoring Carotid Surgery
Acronym: PREST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7539
Record Dates: First submitted 2025-04-04; First posted 2025-04-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Carotid Artery Diseases; Haemodynamic Monitoring
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- predictive (Experimental)
  Interventions: Other: predictive approach to hemodynamic management
- standard (No Intervention): hemodynamic optimization will be made based on a standard protocol

INTERVENTIONS:
Other: predictive approach to hemodynamic management — vasoactive drugs and fluids will be given based on the hypotension prediction index
  Arms: predictive

SUMMARY:
patients scheduled for carotid endoarterectomy will be randomly assigned to a group in which arterial hypotension will be avoided by a predictive haemodynamic approach or to a group in which arterial hypotension will be treated in a standard manner

ELIGIBILITY:
Inclusion Criteria:

- >18 years old patients

Exclusion Criteria:

* Body MassIndex > 35 Kg /m2;
* Atrial Fibrillation
* Urgent surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
stump pressure | during surgery
  we will compare the value of stump pressure between the two groups. the stump pressure will be measured after clamping the common and external carotid vessels

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No